CLINICAL TRIAL: NCT06480292
Title: Effects of Telerehabilitation Exercise Program on Maternal Quality of Life, Fetal and Neonatal Health Outcomes in Women With Gestational Diabetes Mellitus
Brief Title: Telerehabilitation Exercise: Effects on Maternal Quality of Life, Fetal and Neonatal Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ghazal Fatima
Record Dates: First submitted 2024-06-05; First posted 2024-06-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Intervention Model Description: This will be a comparison between two groups; experimental and control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation exercise program (Experimental): This group will receive a structured tele rehabilitation exercise protocol of low to moderate intensity warm up ,aerobic ,resistance and cool down exercises for 3 times a week progressively increased for 8 weeks. along with routine medical care will be provided.
  Interventions: Other: telerehabilitation exercise
- Routine medical care (Active Comparator): The control group will receive routine medical care including oral medication (metformin), dietry precautions and advised to do regular walk for 20-30minutes.
  Interventions: Other: routine medical care

INTERVENTIONS:
Other: telerehabilitation exercise — 5 min warmup will include ankle plantar and dorsiflexion ,trunk side flexion ,shoulder circles ,shoulder ROMS.it will be followed by 5 min aerobics that includes spot marching and side stepping. it will be followed by resistance exercise which will be divided into 3 groups. each group of exercise will be performed one day each. chair squats, arm pulls, seated triceps, biceps curls etc. are included in these resistance exercises. intensity of each exercise will be progressively increased.
  Arms: Telerehabilitation exercise program
Other: routine medical care — The control group will be given routine medical care (including dietary modification, oral anti diabetics (metformin) and advised to do regular walk (20-30min/day).
  Arms: Routine medical care

SUMMARY:
Gestational diabetes mellitus (GDM) occurs when blood sugar levels rise during pregnancy, typically between 24-28 weeks, affecting about 2-18% of all pregnancies. It is a common metabolic disease that can lead to health risks for the mother, fetus, and child, and can negatively impact the mother's quality of life. This study aims to explore how a telerehabilitation exercise program affects the quality of life of mothers with GDM and the health of fetus/neonate.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) significantly impacts maternal quality of life (QoL) and fetal/neonatal health. According to the World Health Organization, quality of life (QOL) is a person's view of their status in life within their culture and value system. Pregnancies with GDM, negatively affect personal, familial, and social life, leading to poorer QOL. GDM causes medical issues for the mother and fetus and harms the mother's psychological well-being, reducing her QOL. Due to the increasing prevalence of GDM and the importance of improving QOL for affected women, this study examines impact of telerehabilitation exercise on quality of life of pregnant women. Awareness about the importance of exercise in managing gestational diabetes mellitus (GDM) is crucial. Regular physical activity can help control blood sugar levels, reduce insulin resistance, and improve overall health for both the mother and fetus leading to better pregnancy outcomes.Telerehabilitation offers convenience, accessibility, and personalized support, allowing patients to exercise from home with continuous healthcare provider monitoring.It is a cost-effective, flexible, and safer alternative to traditional exercise methods, especially beneficial for managing gestational diabetes.

The control group will recieve routine medical care and the experimental group will recieve structured telerehabilitation exercise protocol. The results of both groups will be recorded and compared to assess the effectiveness of using telerehabilitation in the treatment of women with GDM in improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 35 years
* Gestational age between 20-28weeks
* diagnosed with Gestational diabetes mellitus through oral glucose tolerance test (OGTT)
* Primigravida and multigravida
* able to do 6 6-minute walk tests under a severity level of 6 on the Borg scale of breathlessness.
* Patients or caregivers have and able to use an electronic device (PC, tablet or smartphone)
* Who signed informed consent

Exclusion Criteria:

* Previously diagnosed T1DM or T2DM
* High-risk pregnancy conditions contraindicating exercise as per ACOG guidelines
* Patients taking insulin regularly.
* Patients with fetal anomalies diagnosed at 20 th week.
* Multiple gestation (twin or triplets).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
GDMQ-36 for Maternal Quality of Life | changes from baseline to 8th week
  The GDMQ (Gestational Diabetes Mellitus Quality of Life)-36 is a simple, valid, and reliable tool for assessing the quality of life of women with GDM across five domains: Emotional, Physical, Social, Self-Efficacy, and Healthcare. Each domain includes multiple items rated on a 5-point Likert scale (strongly agree to strongly disagree) with a score range of 1 to 5. Domain scores are calculated by summing the responses for each item, and the total GDMQ score is the sum of all domain scores. Higher scores generally indicate better quality of life if the scale is positively oriented. This tool helps identify areas needing intervention and support, offering a comprehensive measure of GDM-related quality of life.

SECONDARY OUTCOMES:
Fetal Health | changes from baseline to 8th week
  Fetal Health measured by fetal obstetric ultrasound and anomaly scan.
Neonatal Health | At the time of delivery
  Neonatal outcome measured by examination and pediatric records.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (2):
- Pakistan (2):
  - Pakistan Railways Hospital, Rawalpindi, Punjab Province
  - AlKhidmat Razi Hospital,Rawalpindi, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No